CLINICAL TRIAL: NCT01774929
Title: Evaluation of Efficacy and Safety of TTS-Fentanyl in Moderate to Severe Pain in Osteoarthritis Patients
Brief Title: An Efficacy and Safety Study of Transdermal Therapeutic System (TTS)-Fentanyl in Participants With Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014536; FENPAI 4053
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-04

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Transdermal Therapeutic System (TTS)-fentanyl; Durogesic
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transdermal Therapeutic System (TTS)-fentanyl (Experimental): TTS-fentanyl patches releasing at the rate of 12.5 microgram per hour for 3 days. The patches will be replaced every 3 days until 30 days.
  Interventions: Drug: TTS-fentanyl

INTERVENTIONS:
Drug: TTS-fentanyl — TTS-fentanyl patches releasing at the rate of 12.5 microgram per hour for 3 days. The patches will be replaced every 3 days until 30 days.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Transdermal Therapeutic System (TTS)-fentanyl patch (transdermal patch containing a drug that is put on the skin so the drug will enter the body through the skin) in participants with moderate (medium level of seriousness) to severe (very serious, life threatening) pain of osteoarthritis (disorder, which is seen mostly in older persons, in which the joints become painful and stiff).

DETAILED DESCRIPTION:
This is an open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving, "unblinded"), single-arm, prospective (study following participants forward in time), study of TTS-fentanyl in participants with moderate to severe pain of osteoarthritis. The study will consist of 2 phases: screening phase up to 7 days before starting the treatment and treatment phase of 30 days. The first patch will be applied by investigator then by participants until 30 days. The dose of TTS-fentanyl can be increased, if needed, by 12.5 microgram per hour until adequate (reasonably good) pain control is achieved and taking into account the daily dose of supplemental paracetamol required by the participant. Other concomitant (given at the same time) analgesics (drug used to control pain) will not be used during this phase. Efficacy with regard to pain control will be recorded principally by the participant through questionnaires in a daily diary. This record will be used to support more detailed assessments at study visits on Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire. Participants' safety will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (lasting a long time) primary osteoarthritis pain for more than 3 months with Visual Analog Scale (VAS) greater than or equal to 5
* Participants having moderate to severe pain (VAS greater than or equal to 5), which was not adequately controlled by weak opioids such as tramadol or codeine at optimal doses (at least 150 milligram [mg] per day for tramadol or 200 mg per day for codeine) for at least 7 consecutive days
* Participants who failed from other treatments such as operation or lack of efficacy of current treatment

Exclusion Criteria:

* Skin disease that prevents the use of the transdermal system or which could affect the absorption of fentanyl or local tolerability
* History or suspicion of alcohol or drug abuse within the past 5 years
* History of cardiac, nervous system or respiratory disease which in the investigator's judgment precludes participation in the study because of the potential for respiratory depression
* Confusion, reduced level of consciousness, or concomitant (given at the same time) psychiatric disorder which, in the opinion of the investigator, could prevent participation in the trial
* Pregnant or breast-feeding female; female participants of child bearing potential without adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd.,Thailand Clinical Trial, Study Director — Janssen-Cilag Ltd.,Thailand
Locations (1):
- Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- Transdermal Therapeutic System (TTS)-Fentanyl: TTS-fentanyl patches releasing at the rate of 12.5 microgram per hour for 3 days. The patches were replaced every 3 days until 30 days.
Period: Overall Study
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl
Started | 35
Completed | 32
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl
Number analyzed (Participants) | 35
Age Continuous [Mean (Standard Deviation); unit: Years] | 66.03 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 1
Pain Intensity Score by Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: Centimeter [cm]] — Assessed by 10 cm of VAS from 0 to 10, where 0 cm=no pain and 10 cm=worse pain.
  Centimeter [cm] | 7.86 (2.02)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Score at Day 15
Description: The pain intensity was assessed by using a 10 centimeter (cm) Visual Analog Scale (VAS) ranging from 0 cm=no pain to 10 cm=worse pain.
Time Frame: Day 15
Population: Intent to treat (ITT) population included all participants who received at least 1 dose of study medication and had at least 1 post baseline efficacy assessment. "N" signifies those participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl
Number analyzed (Participants) | 33
cm | 6.61 (2.93)

2. Primary Outcome: Pain Intensity Score at Day 30
Description: The pain intensity was assessed by using a 10 cm VAS ranging from 0 cm=no pain to 10 cm=worse pain.
Time Frame: Day 30
Population: ITT population included all participants who received at least 1 dose of study medication and had at least 1 post baseline efficacy assessment. "N" signifies those participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl
Number analyzed (Participants) | 33
cm | 6.00 (3.31)

3. Secondary Outcome: Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) Score at Day 15 and Day 30
Description: The WOMAC is a self-administered; participant reported health status questionnaire designed to capture elements of pain, stiffness and physical impairment in participants with osteoarthritis. It consists of 24 questions (5 questions about pain, 2 about stiffness and 17 about physical function) scored on a VAS of 0 to 10 cm (0 cm=no pain to 10 cm=worse pain). Individual question responses are assigned a score of between 0=extreme and 4=none. Maximum scores for each element differ and therefore, scores were normalized. Total normalized score ranges from 0=worst to 100=best.
Time Frame: Baseline, Day 15 and Day 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl
Number analyzed (Participants) | 33
Units on a scale
  Baseline | 17.04 (4.38)
  Day 15 | 14.84 (5.40)
  Day 30 | 13.41 (6.44)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 30
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 23/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transdermal Therapeutic System (TTS)-Fentanyl (N=35)
Vomiting (General disorders) | 2
Nausea (General disorders) | 7
Constipation (General disorders) | 5
Abdominal pain (General disorders) | 1
Dyspepsia (General disorders) | 1
Drowsiness (General disorders) | 7
Headache (General disorders) | 1
Itching (General disorders) | 3
Irritate (General disorders) | 1
Fatigue (General disorders) | 1
Tinnitus (General disorders) | 1
Vertigo (General disorders) | 3
Lacrimation increased (General disorders) | 1
Dysphonia (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator wishes to publish information from the study, a copy of the manuscript must be provided to the Sponsor for review at least 60 days before submission for publication. If requested by the Sponsor, the Investigator will withhold it up to an additional 60 days to allow for filing of a patent application. The Sponsor will not change or suppress the scientific content. For multicenter study, results may not be published before the primary endpoints of a study have been published.